CLINICAL TRIAL: NCT02755610
Title: Check List to Improve Patient Self-care and Product Defect Report in Continuous Ambulatory Peritoneal Dialysis
Acronym: CLIP-SP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CLIP-SP
Record Dates: First submitted 2016-02-09; First posted 2016-04-29 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2023-08

CONDITIONS: End-Stage Kidney Disease; Peritonitis
Keywords: Peritoneal Dialysis; Checklist
MeSH Terms: conditions — Kidney Failure, Chronic; Peritonitis

STUDY DESIGN:
Intervention Model Description: Participants in the Study Arm receive standard care and a paper check list to record product defect information Participants in the Control Arm receive standard care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD Product Check List (Experimental): PD Product Check List was developed based on the 28 routine steps of standard orientation manual for new Thai PD patients. Of these, step 2 (weighting the PD solution bag), step 3 (checking expiration date, volume, glucose concentration, clarity, and color, step 27 (weighting the PD solution bag), and step 28 (recording time, volume, and any abnormality encountered) are relevant to product defect report.
  Interventions: Other: PD Product Check List
- Control (No Intervention): Standard care

INTERVENTIONS:
Other: PD Product Check List — PD Product Check List was developed based on the 28 routine steps of standard orientation manual for new Thai PD patients. Of these, step 2 (weighting the PD solution bag), step 3 (checking expiration date, volume, glucose concentration, clarity, and color, step 27 (weighting the PD solution bag), and step 28 (recording time, volume, and any abnormality encountered) are relevant to product defect report.
  Arms: PD Product Check List

SUMMARY:
Peritoneal Dialysis (PD) has been the main method of treatment for Thai End-Stage Renal Disease (ESRD) patients under the "PD First" policy of the Universal Coverage (UC) scheme. The increased demand has resulted in not only supply chain logistical problems, but also product quality concerns. Peritonitis, the main complication and checklist cause of failure in Continuous Ambulatory Peritoneal Dialysis (CAPD) patients, could be caused by a product defect. This cluster randomized trial will be conducted in 22 randomly selected PD centers in Thailand to assess if a checklist intervention could reduce peritonitis rate and increase the number of checklist product defect report.

DETAILED DESCRIPTION:
Peritoneal Dialysis (PD) has been the main method of treatment for Thai End-Stage Renal Disease (ESRD) patients under the "PD First" policy of the Universal Coverage (UC) scheme. The increased demand has resulted in not only supply chain logistical problems, but also product quality concerns. Peritonitis, the main complication and main cause of failure in CAPD patients, could be caused by a product defect.

PD Product Check List was developed based on the 28 routine steps of standard orientation manual for new Thai PD patients. Of these, step 2 (weighting the PD solution bag), step 3 (checking expiration date, volume, glucose concentration, clarity, and color, step 27 (weighting the PD solution bag), and step 28 (recording time, volume, and any abnormality encountered) are relevant to product defect report.

This cluster randomized trial will be conducted in 22 PD centers (anticipated 20-25 prevalent and 10-15 incidence PD cases per center) to answer the primary research question: is the checklist intervention effective in reducing peritonitis rate? The secondary research questions will also be considered: does the checklist help increase the number of product defect report?

Peritonitis incidence rate is the primary outcome, defined based on the International Society for Peritoneal Dialysis (ISPD) 2010 recommendation. Product defect incidence is the secondary outcome, measured by a number of incidence of product defect reported by the patients. Given no standard definition, a PD solution product will be considered defective if it is expired on the day of use, incorrect glucose concentration, abnormal clarity or color, physical abnormality of the box and/or the bag, or loose connector.

Because of the nature of the intervention, blinding is not possible. Cluster randomization will be performed to allocate 11 PD centers to the study group and the other 11 PD centers to control group. While all subjects will receive standard PD care, subjects in the study group will also receive the checklist plus a 30-minute orientation of how to use the checklist.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients who start peritoneal dialysis not longer than one month and participate in PDOPPS study

Exclusion Criteria:

* ESRD patients who receive only hemodialysis
* ESRD patients who receive emergency peritoneal dialysis
* Illiterate ESRD patients or their caregivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2016-05-02 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Peritonitis Incidence Rate | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Product Defect Incidence | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Krit Pongpirul, MD,MPH,PhD., Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhanakijcharoen P, Sirivongs D, Aruyapitipan S, Chuengsaman P, Lumpaopong A. The "PD First" policy in Thailand: three-years experiences (2008-2011). J Med Assoc Thai. 2011 Sep;94 Suppl 4:S153-61. PMID 22043584
- [Background] Praditpornsilpa K, Lekhyananda S, Premasathian N, Kingwatanakul P, Lumpaopong A, Gojaseni P, Sakulsaengprapha A, Prasithsirikul W, Phakdeekitcharoen B, Lelamali K, Teepprasan T, Aumanaphong C, Leerawat B, Pongpiyadej J, Srangsomvong S, Kanjanabuch T, Eiam-Ong S, Vareesaengthip K, Lumlertkul D. Prevalence trend of renal replacement therapy in Thailand: impact of health economics policy. J Med Assoc Thai. 2011 Sep;94 Suppl 4:S1-6. PMID 22043559
- [Background] Liu FX, Gao X, Inglese G, Chuengsaman P, Pecoits-Filho R, Yu A. A Global Overview of the Impact of Peritoneal Dialysis First or Favored Policies: An Opinion. Perit Dial Int. 2015 Jul-Aug;35(4):406-20. doi: 10.3747/pdi.2013.00204. Epub 2014 Jul 31. PMID 25082840
- [Background] Wong HS, Ong LM, Lim TO, Hooi LS, Morad Z, Ghazalli R, Shaariah W, Lim YN, Ahmad G, Goh BL, Liaw L, Pee S, Lee ML. A randomized, multicenter, open-label trial to determine peritonitis rate, product defect, and technique survival between ANDY-Disc and UltraBag in patients on CAPD. Am J Kidney Dis. 2006 Sep;48(3):464-72. doi: 10.1053/j.ajkd.2006.05.008. PMID 16931220
- [Background] Kanjanabuch T, Chancharoenthana W, Katavetin P, Sritippayawan S, Praditpornsilpa K, Ariyapitipan S, Eiam-Ong S, Dhanakijcharoen P, Lumlertgul D. The incidence of peritoneal dialysis-related infection in Thailand: a nationwide survey. J Med Assoc Thai. 2011 Sep;94 Suppl 4:S7-12. PMID 22043560
- [Background] Amornnimit W, Pongpirul K, Sampatanukul P, Tungsanga K, Tosukhowong P, Kanjanabuch T. Black-stained peritoneal dialysis tubing: a national survey. Perit Dial Int. 2013 Nov-Dec;33(6):704-7. doi: 10.3747/pdi.2012.00167. No abstract available. PMID 24335129
- [Background] Pongpirul K, Pongpirul WA, Kanjanabuch T. Potential causes of black-stained peritoneal dialysis tubing: an analysis from nurse practitioner's prospect. BMC Res Notes. 2014 Jul 6;7:434. doi: 10.1186/1756-0500-7-434. PMID 24997794
- [Background] Treamtrakanpon W, Katavetin P, Yimsangyad K, Keawsinark P, Sanganunttakan S, Pandon S, Buddeewong D, Prakot A, Khumsupo C, Thamsutee N, Yaibuaiam R, Khumwong S, Towannang P, Theerasin Y, Mahatnan N, Eiam-Ong S, Kanjanabuch T. From the "PD First" policy to the innovation in PD care. J Med Assoc Thai. 2011 Sep;94 Suppl 4:S13-8. PMID 22043561
- [Background] Bernardini J, Price V, Figueiredo A; International Society for Peritoneal Dialysis (ISPD) Nursing Liaison Committee. Peritoneal dialysis patient training, 2006. Perit Dial Int. 2006 Nov-Dec;26(6):625-32. No abstract available. PMID 17047225
- [Background] Perl J, Davies SJ, Lambie M, Pisoni RL, McCullough K, Johnson DW, Sloand JA, Prichard S, Kawanishi H, Tentori F, Robinson BM. The Peritoneal Dialysis Outcomes and Practice Patterns Study (PDOPPS): Unifying Efforts to Inform Practice and Improve Global Outcomes in Peritoneal Dialysis. Perit Dial Int. 2016 May-Jun;36(3):297-307. doi: 10.3747/pdi.2014.00288. Epub 2015 Nov 2. PMID 26526049
- [Background] Li PK, Szeto CC, Piraino B, Bernardini J, Figueiredo AE, Gupta A, Johnson DW, Kuijper EJ, Lye WC, Salzer W, Schaefer F, Struijk DG; International Society for Peritoneal Dialysis. Peritoneal dialysis-related infections recommendations: 2010 update. Perit Dial Int. 2010 Jul-Aug;30(4):393-423. doi: 10.3747/pdi.2010.00049. No abstract available. PMID 20628102
- [Background] Vonesh EF. Modelling peritonitis rates and associated risk factors for individuals on continuous ambulatory peritoneal dialysis. Stat Med. 1990 Mar;9(3):263-71. doi: 10.1002/sim.4780090309. PMID 2188325
- See also: The Peritoneal Dialysis Outcomes and Practice Patterns Study — https://www.dopps.org/AboutUs.aspx